CLINICAL TRIAL: NCT00000385
Title: Long-Term Lithium for Aggressive Conduct Disorder
Brief Title: Long-Term Lithium Treatment for Aggressive Conduct Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Richard P. Malone, MD, Drexel University College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R29MH057093 (NIH); R29MH057093 (NIH); DSIR CT-M
Record Dates: First submitted 1999-11-02; First posted 1999-11-03 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Conduct Disorder; Aggression
Keywords: Aggressive conduct disorder; Adolescence; Child; Conduct Disorder; Female; Lithium; Male; Placebos; Conduct Disorder -- *drug therapy; Lithium -- *therapeutic use
MeSH Terms: conditions — Conduct Disorder; Aggression | interventions — Lithium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Lithium 600 mg to 2700 mg per day
  Interventions: Drug: Lithium
- 2 (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lithium — Lithium 600 mg to 2700 mg per day
  Arms: 1
Drug: Placebo — Matching placebo
  Arms: 2

SUMMARY:
This study will examine the long-term effects of lithium used to treat children and adolescents with aggressive conduct disorder (severe aggression).

DETAILED DESCRIPTION:
Psychotherapeutic agents are often administered without sufficient testing to children and adolescents, often on a long-term basis, to reduce aggression. Many pressures, including managed care, will increase the utilization of pharmacotherapy in the outpatient setting to treat serious problems. Lithium is the most promising agent for the treatment of aggression in children and adolescents. However, it has not been shown that lithium is an effective treatment for these patients in the outpatient (non-hospital) setting, or on a long-term basis. The purpose of this study is to examine the long-term effects of lithium used to treat children and adolescents with aggressive conduct disorder (severe aggression).

The proposed study is a two-phased clinical trial of lithium for the treatment of aggression in conduct disorder. Both phases are double-blind and placebo-controlled with randomization and employ a parallel groups design. Phase 1 contains a short-term 8-week controlled trial, with twice as many subjects randomized to lithium as placebo, increasing the pool of potential lithium responders to continue to Phase 2. In Phase 2, lithium responders from Phase 1 enter a 6-month long-term controlled trial. Every attempt is made to define responders to lithium.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females
2. Ages between 9 and 17 years.
3. Conduct disorder according to DSM-IV (As rated on the DICA-IV).
4. The aggression criterion at screening

Exclusion Criteria:

1. Mental Retardation.
2. Pervasive Developmental Disorder(s).
3. Major Depressive Disorder or Dysthymic Disorder.
4. Bipolar Disorder.
5. Psychotic Disorder (including Schizophreniform Disorder and Schizophrenia).
6. Major medical problem such as cardiac, renal, and thyroid diseases, or seizure disorder.
7. History of psychoactive medication in the previous 2 weeks.
8. Current Pregnancy in females.
9. History of Substance Dependence in the past month.
10. Prior to the proposed study, a history of lithium treatment with serum lithium levels of 0.4 mEq/L or higher for a cumulative period of greater than 10 days.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 1997-09; Primary Completion 2003-12 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Overt Aggression Scale-Modified | Weekly in short term phase, Monthly in long-term phase
Clinical Global Impressions-Improvement Item | Weekly in short term phase, Monthly in long-term phase

SECONDARY OUTCOMES:
Children's Psychiatric Rating Scale-Selected Items | Weekly in short term phase, Monthly in long-term phase
IOWA | Weekly in short term phase, Monthly in long-term phase
DOTES | Weekly in short term phase, Monthly in long-term phase
TESS | Weekly in short term phase, Monthly in long-term phase

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Malone, MD, Principal Investigator — Drexel University College of Medicine
Locations (1):
- Drexel University College of Medicine at Friends Hospital, Philadelphia, Pennsylvania, United States